CLINICAL TRIAL: NCT05648877
Title: Role Of Retrograde Intrarenal Surgery In Management Of Renal Stones: Single Center Experience
Brief Title: to Study the Role of Retrograde Intrarenal Surgery in Management of Renal Stones
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Menoufia University (Other)
Responsible Party: Principal Investigator, Mohammed Ali abdelghaffar, Menoufia gevernorate, Menoufia University
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 11/2020 urol
Record Dates: First submitted 2020-10-01; First posted 2022-12-13 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Retrograde Intrarenal Surgery In Management Of Renal Stones
Keywords: Renal pelvic stone; Semi-rigid URS; Flexible URS; Treatment
MeSH Terms: interventions — Ureteroscopes

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 43 semirigid ureteropyeloscopy (Experimental): 43 Patients underwent semirigid ureteropyeloscopy
  Interventions: Device: Ureteroscope
- 34 flexible ureteropyeloscopy (Active Comparator): 34 patients with flexible ureteropyeloscopy
  Interventions: Device: Ureteroscope

INTERVENTIONS:
Device: Ureteroscope — Role Of Retrograde Intrarenal Surgery In Management Of Renal Stones: Single Center Experience

SUMMARY:
Role Of Retrograde Intrarenal Surgery In Management Of Renal Stones: Single Center Experience

DETAILED DESCRIPTION:
With the advancements in endourologic technology, in the last 30 years, renal stone treatment has dramatically changed, and minimally invasive treatments options, such as extracorporeal shock wave lithotripsy (SWL), percutaneous nephrolithotomy (PCNL), mini-PCNL, retrograde intrarenal surgery (RIRS) or laparoscopy, have replaced open surgery.

Although, minimally invasive treatment modalities have an excellent stone fragmentation rate, the clearance of stone fragments may not be immediate and can occur for any time after the intervention.

The European Association of Urology (EAU) guidelines, recommends PCNL for renal stones greater than 2 cm, and SWL is suggested primarily for stones less than 1 cm in size. Although SWL, RIRS and PCNL are all presented as treatment options for renal stones between, which application is a matter of preference.

The treatment modality selection of renal stones usually depends on stone-related factors (location, size, and composition), clinical factors (patient's comorbidities, patient's compliance, solitary kidney, and abnormal anatomy), and technical factors (equipment available for treatment, success rates, possible complications, invasiveness, the need for anesthetics, hospitalization times, and costs).

PCNL can achieve better results but is more invasive, is associated with greater morbidity and complications, and may be reserved for selected circumstances.

Stone clearance following kidney stone treatment is not well defined. For lower pole stones, Sener and colleagues compared RIRS with SWL and reported a stone-free rate of 52.3% with patients treated using RIRS one week after treatment. However after three months, the stone-free rate improved to 100%.

Ureteroscopic lithotripsy has been the most widely applied treatment for urinary tract stones, with high success and low complication rates. The holmium laser has facilitated the disintegration of stones and increased the effectiveness of ureteroscopic lithotripsy.

Improvements in the new generation of flexible ureteroscopes have made retrograde endoscopic ureteroscopy and laser lithotripsy for renal calculi more popular. The overall success rates of retrograde intrarenal surgery have been reported as 75% to 95% for intrarenal stones > 2 cm after the first or second treatment, whereas the major and minor complication rates vary from 1.5% to 12%, which are less frequent than rates in PCNL procedures.

ELIGIBILITY:
Inclusion Criteria:

* All patients with renal stones were eligible for the procedure. Patients with difficult PCNL

Exclusion Criteria:

* Uncorrected coagulopathy Distal obstruction Active urinary tract infection Ureteropelvic junction obstruction Congenital renal anomalies Staghorn stones

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 77 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2023-02-25 (Estimated); Study Completion 2023-04-01 (Estimated)

PRIMARY OUTCOMES:
stone free rates and complications | Up to 6 months
  Stone free rates of both semirigid and flexible URS

CONTACTS AND LOCATIONS:
Locations (1):
- Menoufia faculty of medicine, Shibīn al Kawm, Monufia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
After completing the thesis, I'll share IPD to other researchers
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: October 2022
Access Criteria: Clinical trial.gov